CLINICAL TRIAL: NCT02067208
Title: Reduced Knee Joint Loading With Lateral and Medial Wedge Insoles for Management of Knee Osteoarthritis: a Randomized Controlled Trial
Brief Title: Wedged Insoles for Management of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Natural Sciences and Engineering Research Council, Canada (Other); Alberta Innovates Health Solutions (Other); Killam Trusts (Unknown); New Balance Athletic Shoe, Inc. (Industry)
Responsible Party: Principal Investigator, Ryan Lewinson, MD/PhD Candidate, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23731-01
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Cartilage; Musculoskeletal; Biomechanics; Subtype; Footwear; Orthotics; Joint Loading
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Orthotic Devices

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Waitlist Control (No Intervention): A waitlist control condition, where the participant receives no insole for 3 months. During this 3 month period, the participant will continue to be monitored for outcome variables.
- Experimental wedged insole (Experimental): Either a medially wedged or laterally wedged footwear insole (whichever reduces knee joint mechanical loading more, as determined from subject-specific biomechanical tests), constructed using a 3D printer will be inserted into each participant's shoe. The participant will be asked to utilize this insole as much as possible throughout the day over the course of 3 months.
  Interventions: Device: wedged insole

INTERVENTIONS:
Device: wedged insole — Wedged insoles are designed to reduce frontal plane knee joint mechanical loads during gait. Specifically, they can alter the knee adduction moment during gait - a variable associated with progression of knee osteoarthritis. In the experimental arm of this study, participants will undergo biomechanical gait analysis to identify the wedged insole that reduces the moments the most. The two options are medial wedge, where the medial aspect of the foot is elevated relative to the lateral aspect, and the lateral wedge, where the lateral wedge is elevated relative to the medial aspect.
  Other Names: orthotic
  Arms: Experimental wedged insole

SUMMARY:
Knee osteoarthritis (OA) is commonly treated using laterally wedged insoles. Although these insoles typically reduce knee abduction moments (KAM) - a variable associated with knee osteoarthritis - and thus are believed to be beneficial for OA management, recent research has indicated that in some cases lateral wedge insoles actually increase knee joint loads. In such cases, a medial wedge may be more appropriate.

The purpose of this study is to evaluate the influence of reduced KAMs on pain over 3-months for patients with knee OA. It is hypothesized that pain reduction will be directly related to KAM reduction.

Forty-six participants with knee OA will be recruited to participate. Each will undergo biomechanical gait analysis to determine the wedge type that most greatly reduces knee adduction moments. In addition, each participant will undergo a Dual Energy X-Ray Absorptiometry (DXA) scan to quantify adiposity. Finally, participants will complete a series of questionnaires to evaluate pain, function, physical activity, footwear comfort and injury history. Participants will be randomized into either a wait list control group (no insole) or experimental group (medial or lateral wedged insole), and monitored for 3 months.

Changes to pain, function, comfort and physical activity from baseline to 3 months will be assessed within the control and experimental groups. Regression analyses will be conducted on the experimental group to determine if a relationship exists between reduced KAMs and reduced pain over 3 months. Comparisons will also be made between the control and experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed knee osteoarthritis (using American College of Rheumatology clinical and radiographic criteria)
* Kellgren-Lawrence grade 1, 2, 3 or 4
* Primary symptoms and disease location must be attributed to medial tibiofemoral compartment
* KOOS pain of 75 points or lower (where 0 is worst pain and 100 is no pain)

Exclusion Criteria:

* X-ray older than 2 years
* Viscosupplementation within past 6 months
* Cortisone injection in past 3 months
* Narcotic pain medication within past 3 months
* Use of knee unloading brace interventions in past 2 months
* Recent (past 6 months) knee or neuromuscular injury that could bias pain assessments or gait analysis results
* No KAM reduction with either lateral or medial wedge insole

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
KOOS pain score | baseline, 1-month, 2-months, 3-months
  Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subsection

SECONDARY OUTCOMES:
Adiposity | baseline
  Measured using Dual Energy X-Ray Absorptiometry (DXA) scan
Knee biomechanics | baseline
  Other knee joint mechanical variables assessed using motion analysis (ex. varus thrust, knee adduction impulse).
PASE score | baseline, 1-month, 2-months, 3-months
  Physical Activity Scale for the Elderly (PASE)
UCLA Physical Activity Score | baseline, 1-month, 2-months, 3-months
  Scale evaluating physical activity levels
Knee Adduction Moment | baseline
  Calculated using inverse dynamics
Footwear Comfort | baseline
  Evaluated using 100mm visual analog scale
KOOS subsection and aggregate scores | baseline, 1-month, 2-months, 3-months
  All other KOOS sections (excluding pain, which is primary outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan T Lewinson, BSc, Principal Investigator — University of Calgary; Kelsey HM Collins, BS, Principal Investigator — University of Calgary; Isabelle A Vallerand, BSc, Principal Investigator — University of Calgary; J Preston Wiley, MD, MPE, Principal Investigator — University of Calgary; Linda J Woodhouse, PhD, PT, Principal Investigator — University of Alberta; Raylene A Reimer, PhD, Principal Investigator — University of Calgary; Jay T Worobets, PhD, Principal Investigator — University of Calgary; Walter Herzog, PhD, Principal Investigator — University of Calgary; Darren J Stefanyshyn, PhD, Principal Investigator — University of Calgary
Locations (1):
- Human Performance Laboratory, University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Lewinson RT, Vallerand IA, Collins KH, Wiley JP, Lun VMY, Patel C, Woodhouse LJ, Reimer RA, Worobets JT, Herzog W, Stefanyshyn DJ. Reduced knee adduction moments for management of knee osteoarthritis:: A three month phase I/II randomized controlled trial. Gait Posture. 2016 Oct;50:60-68. doi: 10.1016/j.gaitpost.2016.08.027. Epub 2016 Aug 26. PMID 27580080
- [Derived] Lewinson RT, Collins KH, Vallerand IA, Wiley JP, Woodhouse LJ, Reimer RA, Worobets JT, Herzog W, Stefanyshyn DJ. Reduced knee joint loading with lateral and medial wedge insoles for management of knee osteoarthritis: a protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2014 Dec 3;15:405. doi: 10.1186/1471-2474-15-405. PMID 25467955